CLINICAL TRIAL: NCT06781944
Title: A Multicenter, Open- Label, Randomized, Clinical Trial to Investigate the Efficacy and Safety of OBINOTUZUMAB Versus Cyclophosphamide Combined With Glucocorticoids in Patients With Primary Membranous Nephropathy (Blossom Study)
Brief Title: OBINOTUZUMAB Versus Cyclophosphamide + Glucocorticoids in Primary Membranous Nephropathy(Blossom Study)
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Huashan Hospital (Other)
Responsible Party: Principal Investigator, Chuanming Hao, Professor, Huashan Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ML45515
Record Dates: First submitted 2024-12-15; First posted 2025-01-17 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2025-12

CONDITIONS: Primary Membranous Nephropathy
MeSH Terms: interventions — obinutuzumab; Glucocorticoids

STUDY DESIGN:
Intervention Model Description: Intervention: Intravenous infusion of 1,000 mg obinutuzumab at weeks 0, 2, 24 and 26,Comparator: Cyclical cyclophosphamide and glucocorticoids
  * Methylprednisolone 500 mg iv will be given for 3 consecutive days at the start of month 1,3,5 and followed by prednisone 0.5mg/kg/d (max 40 mg/d) for 27 days.
  * Oral cyclophosphamide will be given for 30 days in month 2, 4, 6.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Obinutuzumab (Experimental): Intravenous infusion of 1,000 mg obinutuzumab at weeks 0, 2, 24 and 26.
  Interventions: Drug: Obinutuzumab
- Comparator (Other): Comparator
  Interventions: Drug: CTX combined with Glucocorticoids

INTERVENTIONS:
Drug: Obinutuzumab — Drug: Obinutuzumab Intravenous infusion of 1,000 mg obinutuzumab at weeks 0, 2, 24 and 26.
  Arms: Obinutuzumab
Drug: CTX combined with Glucocorticoids — Drug: Glucocorticoids Methylprednisolone 500 mg iv will be given for 3 consecutive days at the start of month 1,3,5 and followed by prednisone 0.5mg/kg/d (max 40mg/d) for 27 days.
  Drug: CTX
  Oral cyclophosphamide will be given for 30 days in month 2, 4, 6.
  Arms: Comparator

SUMMARY:
This is a randomized, parallel group, active-controlled, open-label, Phase III study comparing the efficacy and safety of obinutuzumab versus cyclophosphamide combined with glucocorticoids in patients with primary membranous nephropathy (pMN). Approximately 144 patients with pMN who have been diagnosed by biopsy or serum anti-PLA2R antibody will be enrolled.

Intervention: Intravenous infusion of 1,000 mg obinutuzumab at weeks 0, 2, 24 and 26 Comparator: Cyclical cyclophosphamide and glucocorticoids Methylprednisolone 500 mg iv will be given for 3 consecutive days at the start of month 1,3,5 and followed by prednisone 0.5mg/kg/d (max 40 mg/d) for 27 days.

Oral cyclophosphamide will be given for 30 days in month 2, 4, 6.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18～75 years (including 18 and 75)old at the time of signing Informed Consent Form
* pMN patients diagnosed according to renal biopsy (original biopsy needs to include light, immunofluorescence, and electron microscopy) within 5 years or serum anti-PLA2R antibody (≥14 RU/ml )
* 24-hour UPCR ≥ 4 g/g and serum albumin (sALB) < 30 g/L,despite being treated with ACEi and/or ARB for ≥ 6 months prior to screening, or 24-hour UPCR ≥ 5 g/g and sALB < 30 g/L , despite being treated with ACEi and/or ARB for ≥ 3 months prior to screening; or 24-hour UPCR ≥ 8 g/g and sALB < 25 g/L, despite being treated with ACEi and/or ARB for ≥ 1 month prior to screening,.
* eGFR ≥40 mL/min/1.73m2 (CKD-EPI), a renal biopsy is required to exclude renal damage due to other co-morbidities if eGFR <60mL/min/1.73 m2.
* Ability to comply with the study protocol, in the investigator's judgment

Exclusion Criteria:

* Patients with a secondary cause of MN (e.g. hepatitis B, systemic lupus erythematosus, medications, malignancies)
* Type 1 or 2 diabetes mellitus
* eGFR <40 mL/min/1.73m2 (CKD-EPI) or dialysis or kidney transplantation
* Evidence of 50% reduction in proteinuria or serum anti-PLA2R antibody within 6 months prior to screening

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 144 (Estimated)
Dates: Start 2024-10-23 (Actual); Primary Completion 2028-05-31 (Estimated); Study Completion 2028-05-31 (Estimated)

PRIMARY OUTCOMES:
The proportion of patients who achieve overall remission (OR) (Complete remission [CR] or prtial remission[PR]) assessed by 24-hour urinary protein to creatinine ratio at Month 24 | Month 24
  Collect 24-hour urine from patients in the 24th month and measure the 24-hour urinary protein to creatinine ratio (24-hour UPCR) to evaluate the proportion of patients achieving total response (OR) (complete response [CR] or partial response [PR]).

SECONDARY OUTCOMES:
The proportion of patients who achieve overall remission (OR) (Complete remission [CR] or prtial remission[PR]) assessed by 24-hour urinary protein to creatinine ratio at Month 6 | Month 6
  Collect 24-hour urine from patients in the 6th month and measure the 24-hour urinary protein to creatinine ratio (24-hour UPCR) to evaluate the proportion of patients achieving total response (OR) (complete response [CR] or partial response [PR]).
  * CR is defined as a urinary protein-to-creatinine ratio (UPCR) ≤0.3 g/g (24-hour urine).
  * PR is defined as reduction of urinary protein-to-creatinine ratio (UPCR) (24-hour urine) from baseline ≥ 50% ,plus ≤3.5 g/g but >0.3 g/g.
The proportion of patients who achieve overall remission (OR) (Complete remission [CR] or prtial remission[PR]) assessed by 24-hour urinary protein to creatinine ratio at Month 12 | Month 12
  Collect 24-hour urine from patients in the 12th month and perform 24-hour urinary protein to creatinine ratio (24-hour UPCR) testing to evaluate the proportion of patients who achieve OR(Complete remission [CR] or prtial remission[PR]) .
  * CR is defined as a urinary protein-to-creatinine ratio (UPCR) ≤0.3 g/g (24-hour urine)
  * PR is defined as reduction of urinary protein-to-creatinine ratio (UPCR) (24-hour urine) from baseline ≥ 50% ,plus ≤3.5 g/g but >0.3 g/g
The proportion of patients who achieve CR assessed by 24-hour urinary protein to creatinine ratio at Month 12 | Month 12
  Collect 24-hour urine from patients in the 12th month and measure the 24-hour urinary protein to creatinine ratio (24-hour UPCR) to evaluate the proportion of patients achieving CR.
  · CR is defined as a urinary protein-to-creatinine ratio (UPCR) ≤0.3 g/g (24-hour urine).
The proportion of patients who achieve PR assessed by 24-hour urinary protein to creatinine ratio at Month 12 | Month 12
  Collect 24-hour urine from patients in the 12th month and measure the 24-hour urinary protein to creatinine ratio (24-hour UPCR) to evaluate the proportion of patients achieving PR.
  * PR is defined as reduction of urinary protein-to-creatinine ratio (UPCR) (24-hour urine) from baseline ≥ 50% ,plus ≤3.5 g/g but >0.3 g/g.
The proportion of patients who achieve overall remission (OR) (Complete remission [CR] or artial remission[PR]) assessed by 24-hour urinary protein to creatinine ratio at Month 18 | Month 18
  Collect 24-hour urine from patients in the 18th month and perform 24-hour urinary protein to creatinine ratio (24-hour UPCR) testing to evaluate the proportion of patients who achieve OR(Complete remission [CR] or artial remission[PR]) .
  * CR is defined as a urinary protein-to-creatinine ratio (UPCR) ≤0.3 g/g (24-hour urine).
  * PR is defined as reduction of urinary protein-to-creatinine ratio (UPCR) (24-hour urine) from baseline ≥ 50% ,plus ≤3.5 g/g but >0.3 g/g.
The proportion of patients who achieve CR assessed by 24-hour urinary protein to creatinine ratio at Month 18 | Month 18
  Collect 24-hour urine from patients in the 12th month and measure the 24-hour urinary protein to creatinine ratio (24-hour UPCR) to evaluate the proportion of patients achieving CR.
  · CR is defined as a urinary protein-to-creatinine ratio (UPCR) ≤0.3 g/g (24-hour urine).
The proportion of patients who achieve PR assessed by 24-hour urinary protein to creatinine ratio at Month 18 | Month 18
  Collect 24-hour urine from patients in the 18th month and measure the 24-hour urinary protein to creatinine ratio (24-hour UPCR) to evaluate the proportion of patients achieving PR.
  · PR is defined as reduction of urinary protein-to-creatinine ratio (UPCR) (24-hour urine) from baseline ≥ 50% ,plus ≤3.5 g/g but >0.3 g/g.
The proportion of patients who achieve CR assessed by 24-hour urinary protein to creatinine ratio at Month 24 | Month 24
  Collect 24-hour urine from patients in the 12th month and measure the 24-hour urinary protein to creatinine ratio (24-hour UPCR) to evaluate the proportion of patients achieving CR.
  * CR is defined as a urinary protein-to-creatinine ratio (UPCR) ≤0.3 g/g (24-hour urine).

CONTACTS AND LOCATIONS:
Locations (1):
- Huashan Hospital, Fudan University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided
In signing the final protocol, every participating Investigator agrees to keep all information and results concerning the study and the investigational product confidential for as long as the data remain unpublished. The confidentiality obligation applies to all personnel involved at the investigational site.
  In the conduct of this trial 10 centers will be involved. The size of the author list will be dictated by the journal(s) to which the abstract is submitted, but will include Professor Chuan-Ming Hao, the Primary Investigator for the study, as first or corresponding author. Other named authors will be included up to the maximum number allowed by the journal and will be selected based on recruitment at individual sites. If data is to be presented outside the individual institutions involved in the study, the Sponsor and Steering Committee should approve the content.